CLINICAL TRIAL: NCT01630330
Title: The Role of Contact Force Sensing in Electrical Pulmonary Vein Isolation When Conducting Atrial Fibrillation Ablation
Brief Title: Contact Force Sensing Use in Atrial Fibrillation Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012CI002B
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact Force Known (Active Comparator): Ablation with contact force data known
  Interventions: Procedure: Ablation
- Contact Force Not Known (Experimental): Contact Force data unavailable during ablation
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Atrial Fibrillation Ablation with SmartTouch catheter
  Arms: Contact Force Known
Procedure: Ablation — Atrial Fibrillation Ablation with SmartTouch catheter
  Arms: Contact Force Not Known

SUMMARY:
There are multiple important factors which need to be monitored when conducting ablation for atrial fibrillation. The contact between the catheter tip and the inside of the heart wall is now measurable and may improve the effectiveness of catheter ablation for atrial fibrillation patients.

DETAILED DESCRIPTION:
This study compares patients who have this procedure where this contact information is known (unblinded) versus those where the contact information is not known (blinded). The outcome is the rate of acute reconnection at 1 hour after achieving pulmonary vein isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic AF

Exclusion Criteria:

* Recent CVA
* Contraindication to warfarin therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Acute Pulmonary Vein Reconnection | 1 hour post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton & Harefield Hospital NHS Foundation Trust, London, United Kingdom